CLINICAL TRIAL: NCT06585319
Title: Pilot Study of Kitoscell LP (pirfenidone LP) Vs Collagen-polyvinylpyrrolidone As Treatment and Protection in Patients with Moderate to Severe COVID-19
Brief Title: Pirfenidone LP or Collagen-polyvinylpyrrolidone in COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Materno-Perinatal Hospital of the State of Mexico (Other)
Responsible Party: Principal Investigator, Hugo Mendieta Zeron, Clinical Professor, Materno-Perinatal Hospital of the State of Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-12-713
Record Dates: First submitted 2024-09-01; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: COVID 19
Keywords: collagen-polyvinylpyrrolidone; pirfenidone; survival; immunomodulation
MeSH Terms: conditions — COVID-19 | interventions — collagen-PVP; pirfenidone

STUDY DESIGN:
Intervention Model Description: Patients were assigned one of the following treatments: pirfenidone (KitosCell tabs, CellPharma S de RL de CV. Mexico City, Mexico) 1,200 mg of oral q12 h or collagen-PVP (Fibroquel, Aspid SA de CV, Mexico City, Mexico) 2 ml intramuscular q24 h, for 7 days; control group was of patients without pirfenidone or collagen-PVP. Body temperature, heart rate, respiratory rate, pSO2%, PCO2, and pO2, hematic biometry, serum concentrations of glucose, uric acid, cholesterol, and triacyl glycerides, IFN-γ, TNF-α, IL-2, -4, -10, -13 and -17 were measured at the beginning and after 7 days of treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Collagen-polyvinylpyrrolidone (Experimental): Collagen-PVP ml intramuscular q24 h
  Interventions: Drug: Collagen-polyvinylpyrrolidone
- Pirfenidone (Active Comparator): Pirfenidone 1,200 mg of oral q12 h
  Interventions: Drug: Pirfenidone 1200 mg
- Control (No Intervention): Standard treatment with dexamethasone (intravenously) and 40 or 60 mg of enoxaparin (subcutaneously, according to the patient's weight) once daily and 1 g of paracetamol

INTERVENTIONS:
Drug: Collagen-polyvinylpyrrolidone — 2 ml intramuscular q24 h
  Arms: Collagen-polyvinylpyrrolidone
Drug: Pirfenidone 1200 mg — 1,200 mg of oral q12 h
  Arms: Pirfenidone

SUMMARY:
Collagen-polyvinylpyrrolidone (collagen-PVP) and pirfenidone have the ability to control cytokine storms. This work explores the therapeutic effects of both, on the early treatment of patients with severe COVID-19. The hospital stay, quick COVID-19 severity index (qCSI) and admission to the ICU were statistically significantly lower when the patients were treated with collagen-PVP or pirfenidone, compared to the controls treated with dexamethasone alone.

DETAILED DESCRIPTION:
The therapeutic target of COVID-19 is focused on the control of inflammation and the prevention of fibrosis. Collagen-polyvinylpyrrolidone (collagen-PVP) and pirfenidone have the ability to control cytokine storms observed in rheumatic and fibrotic disorders. In this work, the investigators explored the therapeutic effects of both, in addition to dexamethasone, on the early treatment of patients with severe COVID-19. The hospital stay, quick COVID-19 severity index (qCSI) and admission to the ICU were statistically significantly lower when the patients were treated with collagen-PVP or pirfenidone, compared to the controls treated with dexamethasone alone. Furthermore, only collagen-PVP normalized serum glucose at discharge. Since the intracellular mechanism of action of pirfenidone is partially known, it was performed a whole human genome microarray assay with total RNA isolated from fibroblast and macrophage cultures treated with collagen-PVP. Ingenuity Pathway Analysis showed that cell cycle, inflammation, and cell surface-extracellular matrix interaction could be regulated by the collagen-PVP copolymer, by down-regulation of pro-inflammatory cytokines, such as IL-6 and -8, while Th2 anti-inflammatory response signaling could be up-regulated. Additionally, down-regulation of some of the genes involved in nitric oxide production by inducible nitric oxide synthase showed a possible control for JAK, in the IFN-γ pathway, allowing the possibility of controlling inflammation through the JAK/STAT pathway, as has been observed for pirfenidone and other immunomodulators, such as ruxolitinib. In summary, once again, collagen-PVP and pirfenidone have demonstrated to favor inflammatory control and stand out as a possible therapy for inflammatory disorders derived from viral or microorganism infections.

ELIGIBILITY:
Inclusion Criteria:

* patients infected with SARS-CoV-2, hospitalized, with total bilirubin ≤1.5

Exclusion Criteria:

* if the patient underwent treatment with biological antirheumatic drugs, disease modifiers (DMARDs) or other immunosuppressive agents, patients who required continuous therapy with systemic corticosteroids in a dose greater than 10 mg of prednisone per day or equivalent; pregnant women, calculated creatinine clearance (or estimated glomerular filtration rate less than 10 ml/min or patients requiring renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Number of patients that survived the COVID-19 infection | From enrollment until one month of follow up
  After each of the treatments that were given for seven days, the evolution of the patients was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Mendieta Zerón, PhD, Principal Investigator — Mónica Pretelini Sáenz Maternal Perinatal Hospital
Locations (1):
- Monica Pretelini Saenz Maternal Perinatal Hospital, Toluca, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: No
Because patients were treated in COVID Hospitals with restricted access, information could only be shared through a request from institution to institution with a detailed explanation of the reason for the consultation.

REFERENCES:
- [Background] Leyva-Gomez G, Lima E, Krotzsch G, Pacheco-Marin R, Rodriguez-Fuentes N, Quintanar-Guerrero D, Krotzsch E. Physicochemical and functional characterization of the collagen-polyvinylpyrrolidone copolymer. J Phys Chem B. 2014 Aug 7;118(31):9272-83. doi: 10.1021/jp502476x. Epub 2014 Jul 30. PMID 25051159
- [Background] Olmos-Zuniga JR, Silva-Martinez M, Jasso-Victoria R, Baltazares-Lipp M, Hernandez-Jimenez C, Buendia-Roldan I, Jasso-Arenas J, Martinez-Salas A, Calyeca-Gomez J, Guzman-Cedillo AE, Gaxiola-Gaxiola M, Romero-Romero L. Effects of Pirfenidone and Collagen-Polyvinylpyrrolidone on Macroscopic and Microscopic Changes, TGF-beta1 Expression, and Collagen Deposition in an Experimental Model of Tracheal Wound Healing. Biomed Res Int. 2017;2017:6471071. doi: 10.1155/2017/6471071. Epub 2017 May 11. PMID 28584818
- [Background] Furuzawa-Carballeda J, Cabral AR, Zapata-Zuniga M, Alcocer-Varela J. Subcutaneous administration of polymerized-type I collagen for the treatment of patients with rheumatoid arthritis. An open-label pilot trial. J Rheumatol. 2003 Feb;30(2):256-9. PMID 12563677
- [Background] Kinross P, Suetens C, Dias JG, Alexakis L, Wijermans A, Colzani E, Monnet DL; European Centre for Disease Prevention and Control (ECDC) Public Health Emergency Team; ECDC Public Health Emergency Team. Rapidly increasing cumulative incidence of coronavirus disease (COVID-19) in the European Union/European Economic Area and the United Kingdom, 1 January to 15 March 2020. Euro Surveill. 2020 Mar;25(11):2000285. doi: 10.2807/1560-7917.ES.2020.25.11.2000285. Epub 2020 Mar 16. PMID 32186277